CLINICAL TRIAL: NCT07295301
Title: A Clinical Applied Study on the Impact of Different Early Protein Supplementation Levels on the Prognosis of Neurocritical Patients
Brief Title: Protein Intake Dosage on the Prognosis of Neurocritical Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wenshan City People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025AE003
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Neurocritical Conditions; Traumatic Brain Injury; Ischemic Stroke
Keywords: neurocritical care; protein supplementation; Glasgow Coma Scale; randomized controlled trial; ICU; nutrition
MeSH Terms: conditions — Brain Injuries, Traumatic; Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to three parallel groups, each receiving different protein supplementation regimens, with outcomes compared simultaneously.
Who Masked: Outcomes Assessor
Masking Description: Only outcomes assessors (neurophysicians evaluating GCS scores) are masked to group assignments. Participants, care providers, and investigators are not masked. No other parties are masked in this clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low-Dose Protein Supplementation Group (1.0-1.2 g/kg/d) (Experimental): Enteral nutrition is initiated within 48 hours of ICU admission. From day 1 to day 4, protein dosage is 0.2-0.8 g/kg/d, energy is 5-10 kcal/kg/d. From day 5 to day 7, dosage is gradually increased, with protein dosage 0.8-1.0 g/kg/d, energy 15-20 kcal/kg/d. From day 8 to day 14, participants receive protein supplementation at 1.0-1.2 g/kg/d via enteral nutrition. Observation period lasts 14 days.
  Interventions: Dietary Supplement: Low-Dose Enteral Protein Supplementation (Enteral Nutrition Formulas + Whey Protein Powder)
- Moderate-Dose Protein Supplementation Group (1.3-1.5 g/kg/d) (Experimental): Enteral nutrition is initiated within 48 hours of ICU admission. From day 1 to day 4, protein dosage is 0.2-0.8 g/kg/d, energy is 5-10 kcal/kg/d. From day 5 to day 7, dosage is gradually increased, with protein dosage 0.8-1.0 g/kg/d, energy 15-20 kcal/kg/d. From day 8 to day 14, participants receive protein supplementation at 1.3-1.5 g/kg/d via enteral nutrition. Observation period lasts 14 days.
  Interventions: Dietary Supplement: Moderate-Dose Enteral Protein Supplementation (Enteral Nutrition Formulas + Whey Protein Powder)
- High-Dose Protein Supplementation Group (Above 1.6 g/kg/d) (Experimental): Enteral nutrition is initiated within 48 hours of ICU admission. From day 1 to day 4, protein dosage is 0.2-0.8 g/kg/d, energy is 5-10 kcal/kg/d. From day 5 to day 7, dosage is gradually increased, with protein dosage 0.8-1.0 g/kg/d, energy 15-20 kcal/kg/d. From day 8 to day 14, participants receive protein supplementation at above 1.6 g/kg/d via enteral nutrition. Observation period lasts 14 days.
  Interventions: Dietary Supplement: High-Dose Enteral Protein Supplementation (Enteral Nutrition Formulas + Whey Protein Powder)

INTERVENTIONS:
Dietary Supplement: Low-Dose Enteral Protein Supplementation (Enteral Nutrition Formulas + Whey Protein Powder) — This intervention provides enteral protein supplementation for neurocritical patients in the ICU, using enteral nutrition formulas (in powder or emulsion form). When the protein dosage of the enteral nutrition formula is insufficient, whey protein powder is added; intravenous amino acids are used as an alternative only when patients refuse whey protein powder supplementation. The intervention is initiated within 48 hours of ICU admission, with the protein dosage adjusted gradually: 0.2-0.8 g/kg/d from day 1 to day 4, 0.8-1.0 g/kg/d from day 5 to day 7, and then maintained at 1.0-1.2 g/kg/d from day 8 to day 14. It is administered daily via oral intake or tube feeding.
  Arms: Low-Dose Protein Supplementation Group (1.0-1.2 g/kg/d)
Dietary Supplement: Moderate-Dose Enteral Protein Supplementation (Enteral Nutrition Formulas + Whey Protein Powder) — Enteral protein supplementation for neurocritical patients in the ICU, using enteral nutrition formulas (including powders or emulsions). Whey protein powder is added when the protein dosage of the enteral nutrition formula is insufficient. Initiated within 48 hours of ICU admission, with dosage adjusted gradually: 0.2-0.8 g/kg/d from day 1 to day 4, 0.8-1.0 g/kg/d from day 5 to day 7, and then maintained at 1.3-1.5 g/kg/d from day 8 to day 14. Administered via oral intake or tube feeding, daily.
  Arms: Moderate-Dose Protein Supplementation Group (1.3-1.5 g/kg/d)
Dietary Supplement: High-Dose Enteral Protein Supplementation (Enteral Nutrition Formulas + Whey Protein Powder) — Enteral protein supplementation for neurocritical patients in the ICU, using enteral nutrition formulas (including powders or emulsions). Whey protein powder is added when the protein dosage of the enteral nutrition formula is insufficient. Initiated within 48 hours of ICU admission, with dosage adjusted gradually: 0.2-0.8 g/kg/d from day 1 to day 4, 0.8-1.0 g/kg/d from day 5 to day 7, and then maintained at above 1.6 g/kg/d from day 8 to day 14. Administered via oral intake or tube feeding, daily.
  Arms: High-Dose Protein Supplementation Group (Above 1.6 g/kg/d)

SUMMARY:
This study investigates the effect of different early protein supplementation levels (1.0-2.0g/kg/d, divided into three groups) on the prognosis of neurocritical patients, focusing on the 28-day Glasgow Coma Scale (GCS) score improvement rate. Participants will be randomly assigned to receive varying protein doses, and their short-term (28-day mortality, ICU stay, complications) and long-term (90-day mortality, readmission rate) clinical outcomes will also be compared.

DETAILED DESCRIPTION:
This single-center randomized trial enrolls neurocritical patients (e.g., severe brain injury, stroke) who have been in the ICU for ≥72 hours. Participants are randomly assigned to three groups with different early protein supplementation levels (1.0-1.2g/kg/d, 1.3-1.5g/kg/d, ≥1.6g/kg/d) for 14 days. The primary outcome is the 28-day Glasgow Coma Scale (GCS) score improvement rate (defined as GCS ≥13 or an absolute increase of ≥3 points from baseline). We also assess short-term (28-day mortality, ICU/hospital stay, ventilator-associated pneumonia) and long-term (90-day mortality, readmission rate, tracheostomy rate) clinical results. Data will be collected prospectively to find the optimal protein dose for neurocritical patients.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

Age: 18-80 years old. Disease Diagnosis and Hospitalization: Meets any neurocritical disease diagnosis and requires admission to the neurosurgical ICU for ≥72 hours (based on 2022 Consensus on Chinese Neurosurgical Critical Care).

Disease Type (Meet criteria for any one disease):

Severe Acute Ischemic Stroke (AIS): Diagnosed with acute ischemic stroke (sudden neurological deficit like hemiplegia, aphasia, confirmed by CT/MRI) and severe criteria (NIHSS ≥16, large vessel occlusion in internal carotid artery terminal, MCA M1 segment or basilar artery, or ischemic lesion involving >1/3 cerebral hemisphere).

Severe Spontaneous Intracerebral Hemorrhage (ICH): Diagnosed with spontaneous ICH (sudden headache/vomiting/neurological deficit, confirmed by CT) and severe criteria (supratentorial hemorrhage ≥30ml / infratentorial hemorrhage ≥10ml, hemorrhage involving brainstem/diencephalon, or GCS ≤8).

Severe Traumatic Brain Injury (TBI): Diagnosed with TBI (trauma history, CT showing intracranial hematoma/brain contusion/diffuse axonal injury) and severe criteria (GCS 3-8 within 6 hours post-injury, intracranial hematoma ≥20ml (epidural ≥30ml / subdural ≥10ml), or combined brainstem injury).

General Neurocritical Inclusion (Meet at least 1):

Altered consciousness: GCS ≤8 (severe consciousness disorder) or progressive deterioration of consciousness within 24 hours before enrollment (e.g., somnolence→stupor→coma).

Respiratory/circulatory instability: Require non-invasive (BiPAP) or invasive mechanical ventilation, or vasoactive drugs (norepinephrine ≥0.1μg/kg/min) to maintain systolic blood pressure ≥90mmHg, or central respiratory rhythm abnormalities (e.g., Cheyne-Stokes respiration, apnea).

Increased intracranial pressure (ICP): Invasive ICP monitoring shows sustained ICP >25mmHg, or CT/MRI suggests pre-herniation signs (ventricular compression, midline shift >5mm, sulcal effacement).

Severe neurological deficit: Quadriplegia (muscle strength ≤2), swallowing disorder (Watada drinking test ≥IV, high risk of aspiration), status epilepticus (seizure >5 minutes or recurrent seizures >30 minutes without consciousness recovery).

Nutritional Support Timing: Initiate enteral nutrition (EN) within 24-48 hours after ICU admission, and expect EN to last ≥5 days.

Nutritional Risk: NUTRIC score ≥5 (high nutritional risk) or NRS-2002 score ≥3. Informed Consent: Signed by the patient or legal guardian (signed by guardian for comatose patients, confirmed by the patient after condition improvement).

Exclusion Criteria:

* Terminal Diseases: Diagnosed with advanced malignant tumor (life expectancy <3 months), irreversible vegetative state (persistent ≥1 month), or long-term renal replacement therapy (RRT) planned to last >2 weeks before enrollment.

Gastrointestinal Contraindications: Complete intestinal obstruction, massive gastrointestinal bleeding within 24 hours (blood transfusion ≥4U), severe intestinal ischemia, short bowel syndrome (remaining small intestine <100cm).

Metabolic Abnormalities: Congenital urea cycle disorder, severe liver failure (Child-Pugh Class C), allergy to the study's enteral nutrition formula (whey protein/short peptide type), uncontrolled diabetes (fasting blood glucose sustained >13.9mmol/L).

Others: Participating in other clinical studies on nutritional intervention, or patient/family refuses to participate.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-06 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Improvement Rate of Glasgow Coma Scale (GCS) Score at 28 Days | 28 days
  Assesses the proportion of ICU neurocritical patients with significant consciousness improvement at 28 days, defined as GCS score ≥13. Baseline GCS (T0) is measured on the enrollment day after vital signs stabilize (e.g., ICP ≤25mmHg, no persistent seizures). The 28-day GCS (T28) is evaluated within 28±3 days: in-hospital patients are scored by neurologists; discharged patients are scored via outpatient visit or structured telephone interview with family. Patients who die within 28 days or have GCS <13 / GCS increase <3 are defined as "not improved".

SECONDARY OUTCOMES:
28-Day Mortality | 28 days
  Assesses the proportion of ICU neurocritical patients who die within 28 days after enrollment. Death events are confirmed via medical records and follow-up interviews.

OTHER OUTCOMES:
Duration of Mechanical Ventilation | Up to 28 days
  Records the total days of mechanical ventilation (invasive/non-invasive) from initiation to discontinuation in ICU neurocritical patients. Data is extracted from ventilator usage and nursing records.
ncidence of Infection | 14 days
  Evaluates the proportion of ICU neurocritical patients developing new infections (e.g., pneumonia, bloodstream infection) within 28 days, diagnosed via clinical symptoms, laboratory tests, and imaging.
Change in Serum Albumin Level | Baseline and 14 days
  Measures the difference in serum albumin concentration from baseline (enrollment day) to 14 days, reflecting nutritional status. Blood samples are tested in the laboratory.
90-Day Mortality | 90 days
  Assesses the proportion of ICU neurocritical patients who die within 90 days after enrollment. Data is collected via medical records, community follow-up, and family telephone interviews.
90-Day Readmission Rate | 90 days
  Evaluates the proportion of ICU neurocritical patients readmitted to the hospital within 90 days after discharge, due to conditions related to the original neurological critical illness or complications. Data is extracted from hospital admission management systems.